CLINICAL TRIAL: NCT01421823
Title: A Double Blinded Study to Examine the Effect of Alpha Agonist Ointment on Fecal Incontinence in Patients With Idiopathic Fecal Incontinence
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RDD Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RDD 111
Record Dates: First submitted 2011-08-21; First posted 2011-08-23 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Idiopathic Fecal Incontinence
Keywords: Fecal Incontinence; Alpha agonist
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- alpha agonist ointment (Experimental)
  Interventions: Drug: alpha agonist ointment
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: alpha agonist ointment — 2 weeks local treatment with alpha agonist ointment
  Arms: alpha agonist ointment
Drug: Placebo — 2 weeks local treatment with placebo ointment
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect and safety of alpha agonist ointment on fecal incontinence severity in patients with idiopathic fecal incontinence.

DETAILED DESCRIPTION:
This is a double blinded cross over study. Approximately 40 subjects will be participating in this 4 weeks study. A screening visit will be used to determine eligibility for the study. Patients found eligible will receive alpha agonist ointment or placebo ointment for 2 weeks. This will be followed by a second 2 weeks treatment cycle in which:

* patients previously treated with alpha agonist will be treated with placebo.
* patients previously treated with placebo will be treated with alpha agonist.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Male or female subjects 18 to 65 years of age.
* Fecal incontinence score over 8.
* The patient is able to understand the treatment and is willing to comply with the prescribed regimen.

Exclusion Criteria:

- Has a clinically significant history or presence of any of the following conditions:

* Known allergy to the API.
* Porphyria.
* Glaucoma.
* Pregnancy or lactation.
* Active or past history of cardiovascular or cerebrovascular disease including unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, congestive heart failure, or cardiac valve abnormalities;
* Type 1 diabetes mellitus;
* Insulin treated type 2 diabetes mellitus.
* Renal insufficiency.
* Liver insufficiency.
* Malignant disease within 5 years of screening;
* Has hypertension (sitting blood pressure over 140/90 mmHg at screening)
* History of rectal surgery.
* History of HIV, hepatitis B, hepatitis.
* Has used, in the last four weeks, drugs that may affect blood coagulation, such as Aspirin (at a dose above 250 mg/day), Warfarin, Sintrom, Enoxaparin, Nadroparin, Heparin, Clopidogrel, Ticlopidine.
* Use of tricyclic or monoamine-oxidase inhibitors.
* Has upon physical examination a rectal deformation or signs of rectal disease such as fissure, bleeding hemorrhoids, fistula., infection or space occupying lesion.
* Unable to understand the use instruction for the ointment, as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Fecal Incontinence | After 2 weeks of treatment
  number of unwanted/unexpected bowel movements in the time period after use of alpha agonist ointment

CONTACTS AND LOCATIONS:
Overall Officials: Yehiel Ziv, MD, Principal Investigator — RDD Pharma Ltd
Locations (1):
- Proctology Clinic, Asaf Harofe Medical Center, Zrifin, Israel